CLINICAL TRIAL: NCT05749185
Title: Comparison Between the Effectiveness of Ultrasound-Guided High Voltage Pulsed Radiofrequency Versus Standard Voltage Pulsed Radiofrequency for Cervical Nerve Roots in Patients With Refractory Chronic Unilateral Cervical Radicular Pain
Brief Title: High Versus Standard Voltage Pulsed Radiofrequency for Cervical Nerve Roots Injection in Refractory Chronic Unilateral Cervical Radicular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, lecturer of anesthesia and pain medicine, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-247
Record Dates: First submitted 2023-02-09; First posted 2023-03-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Cervical Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group H ( high voltage) radiofrequency (Active Comparator): Group H, involved a high voltage PRF technique, where the voltage started at 65 V and could be adjusted up to 80 V based on patient tolerance. Both protocols involved two cycles of PRF application, with each cycle lasting 240 seconds and comprising alternating periods of current application and deactivation. The pulse rate frequency was set at 2 Hertz (Hz), resulting in two active phases/second (20 milliseconds (ms) of current application followed by 480 ms without stimulation).
  Interventions: Device: radiofrequency high voltage
- Group S ( standard) radiofrequency (Active Comparator): utilized a standard voltage PRF technique, administering PRF at a fixed voltage of 45 volts (V).
  Interventions: Procedure: standard RF

INTERVENTIONS:
Device: radiofrequency high voltage — nvolved a high voltage PRF technique, where the voltage started at 65 V and could be adjusted up to 80 V based on patient tolerance. Both protocols involved two cycles of PRF application, with each cycle lasting 240 seconds and comprising alternating periods of current application and deactivation. The pulse rate frequency was set at 2 Hertz (Hz), resulting in two active phases/second (20 milliseconds (ms) of current application followed by 480 ms without stimulation)
  Arms: Group H ( high voltage) radiofrequency
Procedure: standard RF — A standard voltage PRF technique, administering PRF at a fixed voltage of 45 volts (V)
  Arms: Group S ( standard) radiofrequency

SUMMARY:
The goal of this interventional study is to compare efficacy of either standard versus supra-voltage radiofrequency cervical epidural injection in pain alleviation in population with chronic cervical radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years, both genders.
* American Society of Anesthesiologists (ASA) physical status grades I or II.
* Unilateral cervical radicular pain secondary to cervical disc prolapse affecting single nerve root which was refractory to conventional conservative and physiotherapy measures for 12 weeks or more.
* All candidates received 1 millilitre of 2% lidocaine via an ultrasound-guided diagnostic nerve block and informed at least 50% momentary reduction of their pain.
* Diagnosis was confirmed by cervical MRI and nerve conduction tests.

Exclusion Criteria:

* Refusal to participate.
* Cervical radiculopathy pain recurrence after surgery.
* Previous attempt of radiofrequency ablation.
* Concomitant coagulopathic state ( decompensated liver disease, clopidogrel use) .
* Metastatic lesion in the cervical vertebral column.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
visual analogue score | pre-treatment, 1,3, and 6 month after intervention
  Number of patients with successful pain relief at 6 months post-intervention which is defined as more than or equal 50% reduction in VAS from pre-interventional level
  Vas score ranges from 0 to ten . 0= NO pain.... 1-3= mild pain .... 4-6 = moderate pain ... 6-10= severe untearable pain

SECONDARY OUTCOMES:
Neck disability index | pre-treatment, 1,3 and 6 months after intervention
  1- the impact of treatment on the Neck Disability Index which was evaluated before treatment and at 6 months following treatment
Incidence of procedure related adverse events | 6 hours after the procedure
  cervical epidural hematoma, nerve injury

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Raouf, Al Fayyum, Egypt

REFERENCES:
- [Derived] Alsaeid MA, Algyar MF, Mahmoud AM, Farghaly OS, Salah AG, Raouf MM. Ultrasound-guided high-voltage pulsed radiofrequency versus standard-voltage pulsed radiofrequency in refractory chronic cervical radicular pain randomized clinical trial. J Anesth. 2025 Dec;39(6):929-939. doi: 10.1007/s00540-025-03535-5. Epub 2025 Jul 5. PMID 40617971